CLINICAL TRIAL: NCT01797042
Title: A Comparison of the Metabolic Effects of Fructose, Glucose, High Fructose Corn Syrup and Sucrose at Normal Population Consumed Levels on Liver and Muscle Fatty Infiltration, Insulin Resistance, Glucose, Insulin, Leptin, Ghrelin, Postprandial Triglycerides, LDL Particle Size, Uric Acid and Appetite in Adults Aged 20-60 Years Old
Brief Title: A Comparison of the Metabolic Effects of Fructose, Glucose, High Fructose Corn Syrup and Sucrose at Normal Population Consumed Levels in Adults Aged 20-60 Years Old
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rippe Lifestyle Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20122091
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Obesity
Keywords: Fructose; High fructose corn syrup; Energy regulation; Ectopic fat; Understanding; potential
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fructose 9% (Active Comparator): Sugar sweetened milk consumed in an amount that added sugar provides 9% of calories required for weight maintenance
  Interventions: Behavioral: Dietary Compliance
- Glucose 9% (Active Comparator): Sugar sweetened milk consumed in an amount that added sugar provides 9% of calories required for weight maintenance
  Interventions: Behavioral: Dietary Compliance
- High fructose corn syrup 18% (Active Comparator): Sugar sweetened milk consumed in an amount that added sugar provides 9% of calories required for weight maintenance
  Interventions: Behavioral: Dietary Compliance
- Sucrose 18% (Active Comparator): Sugar sweetened milk consumed in an amount that added sugar provides 9% of calories required for weight maintenance
  Interventions: Behavioral: Dietary Compliance

INTERVENTIONS:
Behavioral: Dietary Compliance — Incorporation of sugar sweetened milk into the usual diet. Instruction on how to account for additional calories provided by sugar sweetened milk Weekly compliance checks

SUMMARY:
The purpose of this study is to investigate the acute and chronic effects of consumption fructose containing sugars and glucose in a real word setting when consumed in a manner and amount typical in the American diet.

DETAILED DESCRIPTION:
Fructose is known to be metabolized differently than the other common monosaccharides. In addition to the well know lipogenic effects, more recent evidence has shown that the acute changes in hormones and metabolic parameters that control appetite and energy regulation when with fructose consumption may promote caloric overconsumption and, in the long-term, weight gain. However, fructose is rarely consumed in isolation, but instead is consumed in combination with other sugars (with glucose in the case of the two most common sources of fructose: high fructose corn syrup (HFCS) and sucrose, or as part of a mixed macronutrient meal. As such, the practical significance of these short-term findings of isolated monosaccharide consumption is limited.

AIM 1: investigate the response to ten weeks of daily consumption of different fructose containing sugars and glucose at typical intake levels on various metabolic parameters and on fat content of the liver and skeletal muscle.

AIM 2: To investigate whether ten weeks of daily consumption changes the acute metabolic response when these sugars are consumed as part as mixed nutrient meals.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) 21.0 -33.0

Exclusion Criteria:

* More than a 3% change in weight within the 3 months prior to enrollment in the study.
* Currently smoking cigarettes
* Currently taking any prescription medication for less than 3 months.
* Currently taking a prescription medication for weight loss (4 week wash out period required).
* Currently taking any over-the-counter weight loss supplement/s (2 week wash out period required).
* History of thyroid disease, but not taking medication or medication dosage changed one or more times over last 6 months.
* Diagnosed with Type I or Type II diabetes or prediabetes.
* Major surgery within three months of enrollment.
* History of heart problems (e.g. angina, bypass surgery, MI, etc.) within three months prior to enrollment.
* Presence of implanted cardiac defibrillator or pacemaker.
* Uncontrolled hypertension/high blood pressure.
* History of a surgical procedure for weight loss at any time.
* Gastrointestinal disorders including chronic malabsorptive conditions, peptic ulcer disease, Crohn's disease, chronic diarrhea or active gallbladder disease.
* History of inflammatory bowel disease
* History of fatty liver
* History or presence of cancer (except for successfully resected basal cell carcinoma of the skin more than 6 months prior to enrollment).
* History of clinically diagnosed eating disorders including anorexia nervosa, bulimia nervosa or binge eating disorder.
* Women who are pregnant, lactating or trying to become pregnant.
* History of alcohol dependency
* Currently consuming >14 alcoholic drinks (1 drink = 12 fl oz beer, 4 fl oz wine or 1.5 fl oz liquor) per week and/or unwilling to limit intake to less than 3 drinks per week during study participation.
* Lactose intolerance
* Known allergy to HFCS, sucrose, fructose or glucose.
* Any clinically significant food allergy
* Participation in another clinical trial within 30 days prior to enrollment.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 366 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Changes in the acute metabolic and hormonal response (glucose, insulin, leptin, active ghrelin, triglycerides, uric acid) | Baseline and 10 weeks
Changes in fat content of skeletal muscle and liver | Baseline and 10 weeks

SECONDARY OUTCOMES:
Change in body mass and body composition | Baseline and 10 weeks
Change in fasting levels of biomarkers associated with obesity (glucose, insulin, C Reactive Protein (CRP), lipid panel) | Baseline and 10 weeks
Change in glucose tolerance | Baseline and 10 weeks
  Measured by the area under the plasma curve for 2 hours after an oral glucose challenge (75g glucose)

CONTACTS AND LOCATIONS:
Overall Officials: James M Rippe, MD, Principal Investigator — Rippe Lifestyle Institute
Locations (1):
- Rippe Lifestyle Institute, Celebration, Florida, United States

REFERENCES:
- [Derived] Angelopoulos TJ, Lowndes J, Sinnett S, Rippe JM. Fructose containing sugars do not raise blood pressure or uric acid at normal levels of human consumption. J Clin Hypertens (Greenwich). 2015 Feb;17(2):87-94. doi: 10.1111/jch.12457. Epub 2014 Dec 15. PMID 25496265